CLINICAL TRIAL: NCT04706182
Title: Neurosensory Outcomes With Platelet-Rich Fibrin and Proximal Segment Grooving in Sagittal Split Osteotomy: A Randomized Clinical Trial
Brief Title: Platelet-rich Fibrin and Grooving for Sagittal Split Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jesse Han (Other)
Responsible Party: Sponsor-Investigator, Jesse Han, Resident: School of Dentistry- Resident, Oral & Maxillofacial Surgery, University of Washington
Organization: University of Washington (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00011198
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Inferior Alveolar Nerve Injury; Nerve Injury; Neurosensory Disorder; Mandibular Nerve Injury
MeSH Terms: conditions — Sensation Disorders; Mandibular Nerve Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined PRF and PSG (Experimental)
  Interventions: Procedure: Platelet-rich fibrin (PRF); Procedure: Proximal segment grooving (PSG)
- Only PRF (Experimental)
  Interventions: Procedure: Platelet-rich fibrin (PRF)
- Only PSG (Experimental)
  Interventions: Procedure: Proximal segment grooving (PSG)
- Control (no treatment) (No Intervention)

INTERVENTIONS:
Procedure: Platelet-rich fibrin (PRF) — Platelet rich fibrin (PRF) serves as a structural reservoir of cytokines such as platelet-derived growth factor (PDGF), transforming growth factor (TGF-b), insulin-like growth factor (IGF), platelet factor 4 (PF4) and vascular endothelial growth factor (VEGF) which aids in healing and preventing infection. PRF will be prepared as recommended by the manufacturer (Intra-Lock International) by centrifuging 20 mL of the subject's venous blood for 12 minutes at 2700 rpm, followed by compression. The fibrin clot will then be applied to the SSO site prior to fixation. The blood draw for the PRF will be performed approximately 15 minutes prior to fixation of the mandible. 20 mL will be drawn for each PRF side treated. The blood venous draw will be from the subject's arm or from an existing intra-venous line.
  Arms: Combined PRF and PSG; Only PRF
Procedure: Proximal segment grooving (PSG) — Proximal segment grooving is a mechanical method to create additional space within the inferior alveolar canal to allow the IAN to rest without compression or trauma. The surgeon uses a round or acrylic bur to cautiously remove any bony spicules, and remove cancellous bone in the proximal mandibular segment. PSG will be done by using an acrylic round bur on a surgical handpiece to remove 3 to 4 mm of cancellous bone where the IAN will passively rest into prior to fixation.
  Arms: Combined PRF and PSG; Only PSG

SUMMARY:
Sagittal split osteotomy (SSO) is a common operation done to move the mandible to correct dentofacial deformities and obstructive sleep apnea (OSA). Inferior alveolar nerve (IAN) injury and associated paresthesia is a well-known negative outcome following SSO, causing temporary or sometimes, permanent numbness in the chin and/or lip. There are limited methods to decrease the occurrence and duration of neurosensory dysfunction. Recent research has shown that platelet-rich fibrin (PRF) aids neurosensory recovery after SSO. Another method to minimize nerve injury is proximal segment grooving (PSG) to create space for the nerve to rest. This grooving method has never been formerly reported. The purpose of this study is to answer the following question: Among patients undergoing bilateral sagittal split osteotomy (BSSO) for dentofacial deformity or OSA, do those who receive PRF with or without PSG, compared to those who do not, have shorter times to functional sensory recovery (FSR) of the IAN? The null hypothesis is that there is no difference among 4 treatment groups and neurosensory outcomes. The specific aims of this proposal are to 1) enroll and randomize subjects who will undergo BSSO for correction of dentofacial deformity or OSA into 4 different treatment groups (PSG with PRF, PSG alone, PRF alone, neither PSG or PRF), 2) measure objective and subjective post-operative nerve function at fixed intervals post-operatively for up to 1 year, 3) compare differences in neurosensory outcomes among treatment groups, and 4) identify other variables that might be associated with differences in neurosensory outcomes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include patients ages 18 and older, male or female, with a diagnosis of dentofacial deformity and/or OSA who will undergo BSSO.

Exclusion Criteria:

Exclusion criteria include patients with a history of previous mandibular surgery and preoperative neurosensory dysfunction of the trigeminal nerve. Other exclusion criteria are patients without capacity to consent for themselves or unable to read the consent form. Subjects who have conditions which may impair healing (such those on bisphosphonates treatments, blood thinners, corticosteroids, chemotherapy, etc.) will be excluded from participation in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional sensory recovery (FSR) | 1 year postoperative
  Adopted by the British Medical Research Council (MRC) scale, the primary outcome will be FSR, as defined as static 2-point discrimination less than 20 mm and superficial pain/tactile sensation without over-reaction on exam. Neurosensory parameters assessed will be Level A: static light touch, brush stroke direction and static 2-point discrimination; Level B: tensile light touch, using von Frey's hairs; and Level C: pinprick sensation (pain) and temperature.

SECONDARY OUTCOMES:
Subjective inferior alveolar nerve (IAN) function | 1 year postoperative
  Subjective IAN function will be measured using a visual analogue scale (VAS) and recorded as a continuous variable from 0-10. A score of 0 will represent anesthesia, 1-9 hypoesthesia and 10 normal.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Han, DDS, MD, Principal Investigator — University of Washington
Locations (1):
- Dale S. Bloomquist, DDS, MS, Seattle, Washington, United States